CLINICAL TRIAL: NCT05367635
Title: A Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of SKB315 for Injection in Patients With Advanced Solid Tumors Expressing Claudin18.2
Brief Title: A Study of SKB315 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKB315-I-01
Record Dates: First submitted 2022-04-21; First posted 2022-05-10 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1a：Dose escalation (Experimental): Eleven dose levels are tentatively planned for Phase 1a
  Interventions: Drug: SKB315 for injection
- Phase 1b: Dose expansion (Experimental): The dose of SKB315 for injection in Phase 1b is selected based on the Phase 1a monotherapy dose escalation study.
  Interventions: Drug: SKB315 for injection
- Phase 1b combination (Experimental): The dose of SKB315 for injection in Phase 1b is selected based on the Phase 1a monotherapy dose escalation study.
  Interventions: Drug: SKB315 for injection; Drug: Drug: Tagitanlimab Drug: Capecitabine

INTERVENTIONS:
Drug: SKB315 for injection — SKB315 for injection is an Antibody Drug Conjugates (ADC) drug targeting Claudin18.2. The strength of SKB315 is 200 mg/vial.
Drug: Drug: Tagitanlimab Drug: Capecitabine
  Arms: Phase 1b combination

SUMMARY:
This is a multicenter, open-label, multiple-dose dose finding and expansion study to evaluate the safety, tolerability, pharmacokinetic(PK) profile, and anti-tumor efficacy of SKB315 for injection in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open-label, multiple-dose dose finding and expansion study to evaluate the safety, tolerability, PK profile, and anti-tumor efficacy of SKB315 for injection in patients with advanced solid tumors.The study is divided into Phase 1a and Phase 1b: Phase 1a is a dose escalation study to determine the maximum tolerated dose(MTD); Phase 1b （monotherapy）is a dose expansion study to conduct preliminary evaluation of anti-tumor efficacy and further evaluation of safety, tolerability, PK, and immunogenicity of SKB315.Phase 1b（combination with Tagitanlimab and Capecitabine） is designed to evaluate the efficacy and safety of SKB315 combination with Tagitanlimab and Capecitabine in CLDN18.2-positive of patients with locally advanced, recurrent, or metastatic gastric and esophagogastric junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

Ia&Ib(monotherapy):1) Male or female patients aged 18 to 80 years (inclusive) at the time of signing the informed consent form (ICF); 2) Patients with histologically and/or cytologically confirmed advanced solid tumors who have failed standard of care, or who have no available standard of care regimen, or who are unqualified for standard of care; 3) Consent to provide archival or fresh tumor tissue slides for immunohistochemistry (IHC) assessment, and advanced solid tumors with Claudin 18.2 expression as determined by IHC; 4) Presence of at least one measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1; 5) Eastern Cooperative Oncology Group (ECOG) score of 0 or 1; 6) Estimated survival ≥ 3 months as judged by the investigator; 7) Adequate organ and bone marrow function (no blood components and cytokines are allowed within 2 weeks prior to the first dose) ; 8) Have recovered to ≤ Grade 1 (according to national cancer institute (NCI) common terminology criteria adverse events (CTCAE) V5.0) from previously treated toxicity prior to the first dose of study treatment; 9) Patients of childbearing potential (male or female) must use effective medical contraception during the study and for 6 months after the end of dosing; 10) Patients voluntarily participate in the study, sign the ICF, and will be able to comply with the protocol-specified visits and relevant procedures.

Phase Ib (combination) Inclusion criteria

1. Age 18 to 80 years old (including boundary values);
2. Histopathologically confirmed unresectable locally advanced, recurrent, or metastatic adenocarcinoma of the gastric and gastroesophageal junction 3 positive CLDN18.2 expression in tumor tissue;

4. ECOG score 0-1; 5. Expected survival ≥3 months; 6. There is at least one measurable lesion that meets the RECIST 1.1 criteria; 7. Adequate bone marrow and organ function

Exclusion Criteria:

Ia&Ib(monotherapy)1) Received other drugs in clinical study, major surgeries, or any other anti-tumor therapies within 4 weeks prior to the first dose of study treatment; 2) Received any previous therapy targeting Claudin18.2; 3) Plan to receive any other anti-tumor therapy during the study; 4) Received strong cytochrome P450 3A4(CYP3A4) inhibitors or inducers within 2 weeks prior to the first dose of study treatment or within 5 half-lives of drug elimination, whichever is longer; 5) Have other malignancies within 5 years prior to signing of ICF; 6) Pregnant or lactating women; 7) Known history of allergy to any component of SKB315 or other monoclonal antibodies (mAbs); 8) Known history of alcohol abuse (consumption of more than 14 units of alcohol per week or drug abuse); 9) Patients with active hepatitis B or hepatitis C; 10) Human immunodeficiency virus (HIV) positive; 11) Active severe digestive disease; 12) History of major cardiovascular diseases 13) Confirmed serious lung disease or lung disease that may impair the respiratory reserve function of the patient as judged by the investigator; 14) History of serious dementia, altered mental status, or any psychiatric disorder; 15) Concomitant or known metastases to brain or central nervous system; 16) Have clinically significant systemic diseases that may adversely affect the safety of the study; 17) Subjects who may have poor compliance with the clinical study or have other factors based on which the investigator considers that the subjects are not appropriate to participate in the study.

Ib(combination)

1. HER2 expression in tumor tissue is positive.
2. Has a history of brain metastases.
3. Additional malignancy within the five years prior to the first administration.
4. Has an active autoimmune disease or a history of autoimmune disease.
5. Received systemic use of corticosteroids or other immunosuppressants for immunosuppressive effects within 14 days prior to the first administration.
6. A history of immunodeficiency, including a positive HIV test; Presence of active hepatitis B or hepatitis C.
7. In the investigator's judgment, the subjects has other factors that could have affected the study results or led to the forced termination of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Dose Limiting Toxicities (DLT) | From data of initial dose until up to 21/28 days for treatment
  Incidence of Dose Limiting Toxicities
Phase 1b: Objective Response Rate (ORR) | Up to 2 years
  The sum of the number of cases with Complete Response (CR) and Partial Response (PR) in all treated tumor patients (CR + PR) divided by the total number of cases.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 2 years
  PFS: Time from start of treatment to progression of disease (PD) or death, whichever occurs first, in patients with tumors.
Duration of Response (DOR) | Up to 2 years
  DOR: Time from the start of the first assessment of CR or PR in tumor patients to PD or death due to any reason.
Overall Survival (OS) | Up to 2 years
  OS: Time from start of treatment to death due to any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ba, Professor, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China